CLINICAL TRIAL: NCT00618384
Title: Phase II Study Evaluating Transarterial Chemoembolization (TACE) in Combination With Sorafenib for the Treatment of Advanced Hepatocellular Carcinoma (HCC)
Brief Title: TACE and Sorafenib for Advanced Hepatocellular Carcinoma (HCC)
Acronym: SOCRATES
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOCRATES-072
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: TACE; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Patients with TACE therapy will be treated with Sorafenib (2 x 400 mg/day) until progressive disease
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — patients get transarterial chemoembolization (TACE) will get film-coated tablets of Sorafenib (2 x 400 mg/day) until progressive disease
  Other Names: Nexavar

SUMMARY:
For patients with advanced HCC not suitable for resection or liver transplantation but without extrahepatic manifestations, local therapy with TACE is regarded as standard treatment. The present study is planned to evaluate the combination of TACE and sorafenib. A combination of TACE with a multitarget inhibitor like sorafenib may further improve the outcome of patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* with histologically confirmed HCC not suitable for resection or liver transplantation
* Patients with measurable disease according to RECIST
* Performance status ECOG 0-2
* Normal organ and bone marrow function (defined)
* Women of childbearing potential must have performed a negative serum pregnancy test
* male or female patients must use an approved contraceptive method during treatment and for 3 months after end of treatment after the end of treatment with study medication
* Written informed consent

Exclusion Criteria:

* Patient is eligible for liver resection or liver transplantation
* Extrahepatic tumor manifestation
* Thrombosis of the portal vein
* > 8 points according to Child Pugh classification
* Prior TACE or RFTA or any other local ablative treatment
* Prior systemic anticancer chemotherapy or radiotherapy for HCC
* Total bilirubin > 4.5 mg/dl
* Life expectancy of less than 12 weeks
* Esophageal varices grade III without prophylactic band ligation
* Cardiac diseases (defined)
* Uncontrolled hypertension
* Known or suspected hyperthyroid state
* Known brain metastasis
* Patients with seizure disorder requiring medication
* History of organ allograft
* Active clinically serious infections > CTCAE grade 2
* Thrombotic or embolic events
* Hemorrhage/bleeding event (defined)
* Acute variceal bleeding
* Therapeutic anticoagulation with vitamin K antagonists (defined)
* Known or suspected allergies to sorafenib, doxorubicin or lipiodol or any agent given in the course of this trial
* Contraindications to the use of sorafenib, doxorubicin or lipiodol
* Previous cancer distinct in primary site or histology from HCC (defined)
* substance abuse
* Participation in another clinical trial with any investigational study drug
* Lactating women
* Incapability to give valid informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-01; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
determination of time to progression (TTP) | every 30 days after administration

SECONDARY OUTCOMES:
adverse events | 3-week-periods

CONTACTS AND LOCATIONS:
Overall Officials: A. Erhardt, PD Dr., Principal Investigator — Department of Gastroenterology, Hepatology and Infectiology University Duesseldorf
Locations (6):
- Germany (6):
  - Universitätsklinikum Tübingen Innere Medizin I, Tübingen, Baden-Wurttemberg
  - Medizinische Universitätsklinik Ulm Innere Medizin I, Ulm, Baden-Wurttemberg
  - Klinikum der Universität Großhardern, Munich, Bavaria
  - Universitätsklinikum Hamburg-Eppendorf Zentrum für Innere Medizin, Hamburg, Hamburg
  - Klinikum der Johann-Goethe-Universität, Frankfurt am Main, Hesse
  - Johannes-Gutenberg-Universität Medizinische Klinik, Mainz, Rhineland-Palatinate

REFERENCES:
- [Derived] Erhardt A, Kolligs F, Dollinger M, Schott E, Wege H, Bitzer M, Gog C, Lammert F, Schuchmann M, Walter C, Blondin D, Ohmann C, Haussinger D. TACE plus sorafenib for the treatment of hepatocellular carcinoma: results of the multicenter, phase II SOCRATES trial. Cancer Chemother Pharmacol. 2014 Nov;74(5):947-54. doi: 10.1007/s00280-014-2568-8. Epub 2014 Aug 31. PMID 25173458